CLINICAL TRIAL: NCT01182597
Title: Oral Versus Intravenous Proton Pump Inhibitor Treatment in High-risk Bleeding Peptic Ulcers After Endoscopic Hemostasis: a Prospective Randomized Comparative Study
Brief Title: Oral Versus IV Proton Pump Inhibitor in High-risk Bleeding Peptic Ulcers After Endoscopic Hemostasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Attending physician, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201003039M
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Peptic Ulcers
Keywords: Oral PPI treatment has similar benefit as proton pump inhibitor infusion in patient with bleeding ulcers after combined endoscopic hemostasis
MeSH Terms: conditions — Peptic Ulcer | interventions — Pantoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV PPI (Active Comparator): Pantoprazole 3.3mg/hr for 72hrs
  Interventions: Drug: Pantoprazole (Pantoloc)
- Oral PPI (Experimental): Lansoprazole (Takepron OD) 30mg PO q12h
  Interventions: Drug: Lansoprazole (Takepron OD)

INTERVENTIONS:
Drug: Pantoprazole (Pantoloc) — Pantoprazole (Pantoloc) 3.3mg/hr for 72hrs
  Arms: IV PPI
Drug: Lansoprazole (Takepron OD) — Lansoprazole (Takepron OD) 30mg q12h PO
  Arms: Oral PPI

SUMMARY:
Endoscopic hemostasis has been documented by a number of clinical studies to be effective in decreasing rebleeding, need for emergency surgery, and hospitalization days. Studies showed adjuvant treatment with proton pump inhibitor (PPI) after initial endoscopic hemostasis reduced recurrent ulcer bleeding. However, the optimal dose and route of adjuvant PPI therapy remains controversial. A recent study demonstrated frequent oral PPI offered similar acid control as currently recommended intravenous infusion PPI did in patients with bleeding ulcers. The investigators hypothesize that an frequent oral PPI treatment has similar benefit as proton pump inhibitor infusion in patient with bleeding ulcers after combined endoscopic hemostasis.

DETAILED DESCRIPTION:
Acute peptic ulcer bleeding remains a therapeutic challenge with significant morbidity and mortality. Endoscopic therapy using various modalities significantly reduces re-bleeding, need for surgery and mortality in patients with peptic ulcer bleeding. Endoscopic therapy achieves successful hemostasis in more than 90% of patients, and re-bleeding occurs in 10-30% of patients. Re-bleeding has an important impact on prognosis. Studies showed adjuvant treatment with proton pump inhibitor (PPI) after initial endoscopic hemostasis reduced recurrent ulcer bleeding. Two consensus documents have endorsed a high-dose PPI regimen (80 mg stat followed by an infusion of 8 mg/h for 72 h). The biologically plausible mechanism of benefit of such a high-dose regimen is to promote clot stability by sustaining the intragastric pH above 6. However, the optimal dose and administration route of proton pump inhibitors (PPI) for the prevention of peptic ulcer rebleeding remains unclear.

The use of IV PPIs adds significantly to the cost of patient care in hospital. Recent studies reported oral PPI may have similar acid suppressive effect as high dose PPI infusion. A prospective trial and a retrospective analysis have shown that oral PPI therapy may also be effective in decreasing rebleeding rates in patients with acute gastrointestinal bleeding due to high-risk peptic ulcer disease, and the magnitude of benefit appears similar to what has been demonstrated with IV PPIs. A meta-analysis reported no difference in the magnitude of risk reduction between the oral- and the intravenous-route. Given the significant cost savings over their IV counterparts, oral PPIs would be an attractive choice of therapy in this situation provided that they have a similar efficacy to IV PPIs. However, no studies have directly compared oral and IV PPI therapy in this setting.

We conducted a head-to-head study, comparing two strategies for PPI administration in the prevention of rebleeding, surgery, and death in patients with high-risk bleeding peptic ulcers in whom successful endoscopic hemostasis was achieved.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Confirmed ulcer bleeding with Forrest Ia, Ib, IIa
* Endoscopic hemostasis achieved by combined endoscopic hemostasis
* Informed consent obtained

Exclusion Criteria:

* No consent
* Unsuccessful endoscopic treatment
* Upper GI malignancy
* History of subtotal gastrectomy
* Bleeding tendency, platelet count < 80x109/L, prothrombin time INR >1.5
* Myocardial infarction or cerebrovascular accident within one week
* Ulcer bleeding because of mechanical factors (such as, induction of NG tube)
* Malignancy or other advanced disease with a life expectancy of < 6 months
* IV PPI > 40mg within 24hrs before enrollment
* Decompensated liver cirrhosis
* Requiring dialysis
* Pregnant or lactating women
* History of allergy or severe side effects to lansoparzole or pantoprazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Clinical rebleeding | 30 days
  Clinical rebleeding defines:
  1. Hematemesis, fresh blood in the NG tube aspirate
  2. Hematochezia/melena after a normal stool
  3. Decrease in Hb >= 2 g/dL or an increase in Hb < 1 g/dL during 24 hrs, despite >=2 units of blood transfused during 24 hours
  4. SBP <= 90 mm Hg or HR >= 110 beats/min AND melena/hematemesis

SECONDARY OUTCOMES:
Blood transfusion | 30 day
Need of surgery | 30 days
Lengths of hospital stay | 30 days
Mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Chang Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan Univeristy Hospital Yunlin Branch, Douliu, Taiwan
  - National Taiwan Univeristy Hospital, Taipei, Taiwan